CLINICAL TRIAL: NCT02103153
Title: Clinical Evaluation of the Picosure Laser for the Treatment of Unwanted Tattoos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-PICO532-RG5
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Unwanted Tattoos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Picosure Laser System (Experimental)
  Interventions: Device: Picosure Laser System

INTERVENTIONS:
Device: Picosure Laser System

SUMMARY:
The purpose of this study is to evaluate the PICOSURE Laser System for the treatment of unwanted tattoos

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy non-smoking (must have quit 6 months prior) male or female between 18 and 65 years old.
2. Is willing to consent to participate in the study.
3. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits
4. Has unwanted non-cosmetic tattoo containing red ink, that has not previously been treated, and wishes to undergo laser treatment

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject is hypersensitive to light exposure OR takes photo sensitized medication.
3. The subject has active or localized systemic infections.
4. The subject has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy {greater than 81 mg per day}).
5. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. The subject has used Accutane within 6 months prior to enrollment.
8. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. The subject has a history of keloids.
11. The subject has evidence of compromised wound healing.
12. The subject has a history of basal cell carcinoma, squamous cell carcinoma or melanoma.
13. The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications or has an autoimmune disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Laser & Skin Surgery Center of New York, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Picosure Laser System: Subjects will be treated with 1064nm, 532nm, or 755nm in combination or individually, depending on the color of the tattoo and the skin type of the subject. Since the purpose of the study is to test the overall clearance of the tattoo, breaking the results down by wavelengths is extraneous information. The primary purpose of the study is not to compare the wavelengths against each other, but rather, to examine the overall clearance created by the Picosure Laser System. Furthermore, each wavelength is designed to target a specific color, so a multi-colored tattoo will have a variety of wavelengths used (in combination and individually), all for the primary objective of indicating overall tattoo clearance.
Period: Overall Study
Arm/Group | Picosure Laser System
Started | 44
Completed | 27
Not Completed | 17

BASELINE CHARACTERISTICS:
Groups:
- Picosure Laser System: Picosure Laser System
Arm/Group | Picosure Laser System
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 27
  Race/Ethnicity: Asian | 1
  Race/Ethnicity: African American | 1
  Race/Ethnicity: Hispanic | 9
  Race/Ethnicity: Multiple | 6
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Score I | 4
    Fitzpatrick Skin Score II | 13
    Fitzpatrick Skin Score III | 18
    Fitzpatrick Skin Score IV | 8
    Fitzpatrick Skin Score V | 0
    Fitzpatrick Skin Score VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Tattoo Clearance Percentage Using a Photographic Scale
Description: Clearance will be measured using a clearance aesthetic improvement scale. This scale ranges from 0% to 100%, where 0% is 0% tattoo cleared compared to the baseline tattoo, and 100% is 100% of tattoo cleared compared to the baseline tattoo.
Time Frame: 1-3 month follow up post each subject's last treatment, an average of 17.5 months
Population: 12 subjects were lost to follow up, and 5 subjects withdrew consent.
Measure: Mean (Standard Deviation); unit: percentage of clearance
Units Other Than Participants: tattoos
Groups:
- Picosure Laser System: Picosure Laser System, using a combination of combination or individual frequencies of 532 nm, 755 nm, or 1064 nm.
Arm/Group | Picosure Laser System
Number analyzed (Participants) | 27
Number analyzed (tattoos) | 34
percentage of clearance | 84.7 (16.9)

2. Secondary Outcome: Investigator Satisfaction
Description: Questionnaires were used to assess Investigator satisfaction at the post last treatment follow up visit with their cosmetic results when compared to baseline photos using a four point scale ranging from "extremely satisfied" (3) to "extremely dissatisfied" (0).
Time Frame: Baseline and 2 months post last treatment follow up (+/- 1 month)
Population: 12 subjects were lost to follow up, and 5 subjects withdrew consent.
Measure: Count of Units; unit: tattoos
Units Other Than Participants: tattoos
Groups:
- Picosure Laser System: Subjects will be treated with 1064nm, 532nm, or 755nm in combination or individually, depending on the color of the tattoo and the skin type of the subject. Each wavelength is designed to target a specific color, so a multi-colored tattoo will have a variety of wavelengths used (in combination and individually), all for the primary objective of indicating overall tattoo clearance.
Arm/Group | Picosure Laser System
Number analyzed (Participants) | 27
Number analyzed (tattoos) | 34
tattoos
  Number of Tattoo Results Investigator Was Extremely Dissatisfied With | 0
  Number of Tattoo Results Investigator Was Dissatisfied With | 1
  Number of Tattoo Results Investigator Was Satisfied With | 19
  Number of Tattoo Results Investigator Was Extremely Satisfied With | 14

3. Secondary Outcome: Subject Satisfaction
Description: Questionnaires were used to assess Subject satisfaction at the post last treatment follow up visit with their cosmetic results when compared to baseline photos using a four point scale ranging from "extremely satisfied" (3) to "extremely dissatisfied" (0).
Time Frame: Baseline and 2 months post last treatment follow up (+/- 1 month)
Population: 12 subjects were lost to follow up, and 5 subjects withdrew consent.
Measure: Count of Units; unit: tattoos
Units Other Than Participants: tattoos
Arm/Group | Picosure Laser System
Number analyzed (Participants) | 27
Number analyzed (tattoos) | 34
tattoos
  Number of Tattoo Subjects Were Extremely Dissatisfied With | 1
  Number of Tattoo Subjects Were Dissatisfied With | 5
  Number of Tattoo Subjects Were Satisfied With | 17
  Number of Tattoo Subjects Were Extremely Satisfied With | 11

ADVERSE EVENTS:
Time Frame: Adverse Events occurring will be captured and followed throughout the patients' participation in the study, approximately 23 months.
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Groups:
- Picosure Laser System- 532 nm Wavelength: Picosure Laser System, using a frequency of 532 nm
- Picosure Laser System- 755 nm Wavelength: Picosure Laser System, using a frequency of 755 nm
- Picosure Laser System- 1064 nm Wavelength: Picosure Laser System, using a frequency of 1064 nm
Arm/Group | Picosure Laser System- 532 nm Wavelength | Picosure Laser System- 755 nm Wavelength | Picosure Laser System- 1064 nm Wavelength
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/41
Other Adverse Events (participants affected / at risk) | 27/27 | 27/27 | 41/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Picosure Laser System- 532 nm Wavelength (N=27) | Picosure Laser System- 755 nm Wavelength (N=27) | Picosure Laser System- 1064 nm Wavelength (N=41)
Pain (Nervous system disorders) | 23 | 21 | 31
Erythema (Skin and subcutaneous tissue disorders) | 27 | 27 | 41
Pinpoint Bleeding (Skin and subcutaneous tissue disorders) | 20 | 22 | 23
Edema (Skin and subcutaneous tissue disorders) | 23 | 24 | 34
Crusting (Skin and subcutaneous tissue disorders) | 16 | 14 | 20
Scabbing (Skin and subcutaneous tissue disorders) | 26 | 26 | 38
Blistering (Skin and subcutaneous tissue disorders) | 22 | 21 | 32
Hypopigmentation (Skin and subcutaneous tissue disorders) | 6 | 6 | 8
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 3 | 5
Itching (Skin and subcutaneous tissue disorders) | 8 | 5 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.